CLINICAL TRIAL: NCT02468427
Title: Objective Structured Assessment of Technical Skills (OSATS) Evaluation of Operative-Vaginal Delivery by Vacuum Extraction on a Pelvic Training Model
Brief Title: Objective Structured Assessment of Technical Skills (OSATS) Evaluation of Delivery by Vacuum Extraction
Acronym: VAC-OSATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Clemens Tempfer, Prof. Clemens Tempfer, MD, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VACUUM-OSATS
Record Dates: First submitted 2015-05-03; First posted 2015-06-10 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hands-on Teaching (Experimental): Medical students receive a 30 minutes hands-on training session. All study probands perform assisted delivery (operative vaginal delivery) by vacuum extraction on a pelvic model immediately after the training.
  Interventions: Other: hands-on teaching
- Frontal teaching (Active Comparator): Medical students receive a 30 minutes frontal teaching session using a training video demonstrating how to perform assisted delivery (operative vaginal delivery) by vacuum extraction on a pelvic model immediately after the training.
  Interventions: Other: Frontal teaching

INTERVENTIONS:
Other: hands-on teaching — Training session of 30 minutes duration with every proband performing a vacuum extraction on a pelvic training model.
  Arms: hands-on Teaching
Other: Frontal teaching — Training session of 30 minutes duration consisting of a video which demonstrates how to perform a vacuum extraction on a pelvic training model.
  Arms: Frontal teaching

SUMMARY:
In a prospective, randomized Trial, the investigators compare Hands-on teaching and frontal teaching using a Training Video for learning how to perform an assisted delivery by vacuum extraction on a pelvic Training model. Objective Structured Assessment of Technical Skills (OSATS) scores are the primary outcome. The investigators hypothesize that Hands-on Training is superior to a video-teaching with regard to the OSATS scores achieved by the Trainees.

DETAILED DESCRIPTION:
The optimal mode of Training surgical novices how to perform an assisted delivery by means of vacuum extraction is unknown. We prospectively randomize probands to a 30 min hands-on (group 1) and a 30 min demonstration (group 2) training session teaching a standardized vacuum Extraction (VE) algorithm scheme on a pelvic training model. Probands are tested with a 24 item Objective Structured Assessment of Technical Skills (OSATS) scoring system after training and 48 hours, and 72 hours thereafter. OSATS scores are the primary outcome. Performance time (PT), self assessment (SA), confidence (CON), and global rating scale (GRS) are the secondary outcomes. Statistics will beperformed using Mann-Whitney U-test, chi-square test, and multivariable logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Medical Student
* no previous experience in assisted delivery
* no previous gynecologic surgery training

Exclusion Criteria:

* language barrier
* unwillingness to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
OSATS scores | 5 min after the training
  24 predefined OSATS items

SECONDARY OUTCOMES:
OSATS scores after 48 hours | 48 hours after the training
  24 predefined OSATS items
OSATS scores after 72 hours | 72 hours after the training
  24 predefined OSATS items

CONTACTS AND LOCATIONS:
Overall Officials: Clemens B Tempfer, MD, Principal Investigator — Ruhr University Bochum
Locations (1):
- Dept. OBGYN Ruhr University Bochum, Herne, Germany

REFERENCES:
- [Result] Hilal Z, Kumpernatz AK, Rezniczek GA, Cetin C, Tempfer-Bentz EK, Tempfer CB. A randomized comparison of video demonstration versus hands-on training of medical students for vacuum delivery using Objective Structured Assessment of Technical Skills (OSATS). Medicine (Baltimore). 2017 Mar;96(11):e6355. doi: 10.1097/MD.0000000000006355. PMID 28296771